CLINICAL TRIAL: NCT00789932
Title: Cognitive Behavioral Therapy for Core Autism Symptoms in School-Aged Children: A Randomized, Controlled Trial
Acronym: BIACA-2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Organization for Autism Research (Other)
Responsible Party: Principal Investigator, Jeffrey J. Wood, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OAR-UCLA-2009
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- CBT (Experimental)
  Interventions: Behavioral: cognitive behavioral therapy
- Usual Care (Active Comparator)
  Interventions: Behavioral: Usual community care

INTERVENTIONS:
Behavioral: cognitive behavioral therapy — 32 weeks of CBT, 1.5 hours weekly.
  Arms: CBT
Behavioral: Usual community care — 16 weeks of community care, 16 weeks of CBT, 1.5 hours/week.
  Arms: Usual Care

SUMMARY:
This study is designed to examine the efficacy of a cognitive behavioral therapy (CBT) program for treating core autism symptoms, social and emotional problems, and adaptive behavior deficits in children with autism spectrum disorders.

ELIGIBILITY:
Inclusion criteria:

* 7 - 11 years of age
* meet research criteria for a diagnosis of autism, Asperger Syndrome, or PDD-NOS
* meet DSM-IV criteria for one of the following anxiety disorders: Separation Anxiety Disorder, Social Phobia, Obsessive-Compulsive Disorder
* If taking medication, have maintained a stable dose for 1 month prior to baseline assessment

Exclusion Criteria:

* child has an IQ of less than 80
* begin taking new medication(s) or current medication dose changes either (1) less than 1 month prior to baseline assessment, or (2) during the study period
* for any reason the child or parents appear unable to participate in the treatment program

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2008-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
ADIS-C/P (Anxiety Disorder Interview Schedule for Children and Parents) | 8 months (post-treatment)

SECONDARY OUTCOMES:
Behavioral observations of social responsiveness | 8 months (post-treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Wood, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States